CLINICAL TRIAL: NCT01958359
Title: Screening and Brief Intervention Via IVR for Problematic Use of Alcohol: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/1437-31/4
Record Dates: First submitted 2013-10-06; First posted 2013-10-09 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Problem Drinking
Keywords: Randomized Controlled Trial; Alcohol; Telephone; Mobile phone; Screening; Brief intervention; IVR-based conversation menu with exercises and vignettes
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Short IVR (Experimental): IVR-based alcohol diary with feedback
  Interventions: Behavioral: Short IVR
- Therapeutic IVR (Experimental): IVR-based conversation offering a menu of exercises and vignettes.
  Interventions: Behavioral: Therapeutic IVR
- Control (No Intervention): Untreated control group

INTERVENTIONS:
Behavioral: Short IVR — IVR-based alcohol diary with feedback
  Arms: Short IVR
Behavioral: Therapeutic IVR — IVR-based conversation offering a menu of exercises and vignettes.
  Arms: Therapeutic IVR

SUMMARY:
Objectives: The study evaluates the efficacy of two automated telephony, also known as, Interactive Voice Recognition (IVR) interventions, Short IVR and Therapeutic IVR. The Short IVR works as an interactive alcohol diary where the user is contacted once a week for four weeks to register their alcohol consumption during the preceding week. The user is given feedback on changes in alcohol consumption compared to last week. The Therapeutic IVR contacts the user once a week for four weeks and is also available for user-initiated calls 24/7 during this four-week period. The Therapeutic IVR allows the user to traverse a menu where the user chooses among listening to vignettes and doing exercises with the purpose of looking at alcohol consumption and exploring ways of coping with it.

Method: The design is a three-armed randomized controlled design, and outcomes are measured in terms of changes in problematic alcohol use at follow up six months after study initiation and baseline data gathering. Participants with problematic alcohol use (AUDIT >7 for men and >5 for women) are randomized into one of three groups: 1. Short IVR, 2. Therapeutic IVR and 3. Control group. Outcomes on alcohol use as well as information on the users' satisfaction with the intervention are assessed after 6 months.

The primary hypothesis for this study is that having access to one of the two IVR interventions will lead to a greater reduction of problematic alcohol use compared to controls who undergo only screening and follow-up assessment. The secondary hypothesis is that having access to either Short IVR or Therapeutic IVR leads to comparable reductions in risky drinking.

ELIGIBILITY:
Inclusion Criteria:

* AUDIT >7 for men or AUDIT >5 for women.

Exclusion Criteria:

* AUDIT <8 (men) or <6 (women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
AUDIT | 6 months
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems).

SECONDARY OUTCOMES:
User satisfaction | 6 months
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems).

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Department of Clinical Neuroscience, Stockholm, Sweden

REFERENCES:
- [Derived] Andersson C, Gajecki M, Ojehagen A, Berman AH. Automated telephone interventions for problematic alcohol use in clinical and population samples: a randomized controlled trial. BMC Res Notes. 2017 Nov 28;10(1):624. doi: 10.1186/s13104-017-2955-4. PMID 29183357
- See also: Study information site. — http://www.telecoach.eu